CLINICAL TRIAL: NCT01617980
Title: Multimodal Hypoxia Imaging and Intensity Modulated Radiotherapy for Inoperable Non-small-cell Lung Cancer
Acronym: HIL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: German Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HIL-DOT-MOBI
Record Dates: First submitted 2012-04-10; First posted 2012-06-13 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Hypoxia imaging; FMISO-PET; functional MRI; Intensity modulated radiation therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Multimodal hypoxia imaging (Other): Patients with inoperable, stage III non-small cell lung cancer receive serial 18F-FMISO dPET-CT and functional MRI investigations prior, during and post radiation treatment
  Interventions: Other: Multimodal hypoxia imaging

INTERVENTIONS:
Other: Multimodal hypoxia imaging — Patients with inoperable, stage III non-small cell lung cancer receive serial 18F-FMISO dPET-CT and functional MRI investigations prior, during and post radiation treatment

SUMMARY:
Radiotherapy, preferably combined with chemotherapy, is the treatment standard for locally advanced, unresectable non-small cell lung cancer (NSCLC). The tumor response to different therapy protocols is variable, with hypoxia known to be a major factor that negatively influences treatment effectiveness. Visualisation of tumor hypoxia prior to the use of modern radiation therapy strategies, such as intensity modulated radiation therapy (IMRT), might allow higher dose applications to the target volume, leading to improvement of therapy outcome. 18F-fluoromisonidazole dynamic positron emission tomography and computed tomography (18F-FMISO dPET-CT) and functional magnetic resonance imaging (functional MRI) are attractive strategies for imaging tumor hypoxia. The HIL trial is a single centre pilot study combining multimodal hypoxia imaging with 18F-FMISO dPET-CT and functional MRI and intensity modulated radiation therapy (IMRT) in patients with inoperable stage III NSCLC. 15 patients are recruited in the study. All patients undergo serial 18F-FMISO dPET-CT and functional MRI before treatment, at week 5 of radiotherapy and 6 weeks post treatment. Radiation therapy is performed as inversely planned IMRT after four dimensional computed tomography (4D-CT) based target volume definition. Hypoxia imaging is not included in target volume definition or IMRT dose prescription.

Objectives of the trial are to characterize the correlation of 18F-FMISO dPET-CT and functional MRI for tumor hypoxia imaging in NSCLC and evaluate possible effects of radiation therapy on tumor re-oxygenation. Further objectives include the generation of data regarding the prognostic value of 18F-FMISO dPET-CT and functional MRI for locoregional control, progression free survival and overall survival of NSCLC treated with IMRT, which will form the basis for larger clinical trials focusing on possible interactions between tumor oxygenation and radiation outcome.

DETAILED DESCRIPTION:
The HIL-trial has been designed by the study initiators at the Clinical Cooperation Unit Radiation Oncology at the German Cancer Research Center (DKFZ), the Clinical Cooperation Unit Nuclear Medicine at DKFZ, the Department of Radiology at DKFZ and the Department of Radiation Oncology at the University Clinic Heidelberg. The trial is carried out at DKFZ in co-operation with the Department of Radiation Oncology at the University Clinic Heidelberg.

Aim of the study is to characterize the correlation of 18F-FMISO dPET-CT and functional MRI for tumor hypoxia imaging in patients with stage III NSCLC, treated with intensity modulated radiotherapy (IMRT) and evaluate changes in tumor oxygenation during radiation treatment. Objectives include the evaluation of the prognostic value of multimodal hypoxia imaging for locoregional control, progression free survival and overall survival of patients with NSCLC treated with IMRT.

The study is designed as a single centre pilot trial with an accrual of 15 patients with inoperable stage III NSCLC. Patients fulfilling the inclusion criteria are treated with intensity modulated radiation therapy (IMRT). All patients undergo serial 18F-FMISO dPET-CT and functional MRI before treatment, at week 5 of radiotherapy and 6 weeks post treatment.

Eligible patients are informed about participation in the trial with possible benefits and risks, and written informed consent is obtained. Staging is completed through performance of thoracic CT scan, abdominal ultrasound and 18F-FDG dPET-CT scan.

After immobilization in a vacuum mattress a contrast-enhanced thoracic CT scan including four dimensional respiratory triggering is carried out. CT data are synchronized with the recorded respiratory signal and four-dimensional reconstructions are performed to evaluate the motion of the thoracic organs and the tumor during the breathing cycle. Based on the 4D-CT data set, radiation treatment planning is carried out as inverse planning.

Radiation therapy is performed as intensity modulated radiation therapy (IMRT). A dose of 50-54 Gy is applied to the primary tumor and mediastinal lymph nodes in daily fractions of 5 × 2 Gy. Subsequently, the primary tumor and involved lymph nodes are boosted to a total dose of 60-72 Gy in daily fractions of 5 × 2 Gy. Tolerance doses of thoracic organs at risk are not exceeded.

Treatment is carried out on an out-patient basis unless the condition of the patient requires hospital administration.

18F-FMISO is provided by Iason (Graz, Austria). 18F-FMISO dPET-CT investigations are performed prior to radiotherapy, at week 5 of radiation therapy and at 6 weeks post treatment. dPET-CT examinations are performed after the i.v. injection of 18F-FMISO using an Biograph mCT S128(Siemens Medical Solutions Co., Erlangen, Germany). The dynamic studies are acquired with a 28-frame protocol for one hour. Quantification is performed following the iterative reconstruction of the dPET-CT data using a dedicated software package. Generally, volumes-of-interest (VOIs) are placed over the tumor and reference regions, followed by a compartment and non-compartment analysis. A two-tissue compartment model is the model of choice and five parameters will be obtained. The quantification includes the calculation of the fractional blood volume, also named as vessel density (VB), the parameters k1 and k2, which reflect the influx and efflux of FMISO into and out of the cells, and k3 and k4, which are related to the trapping and re-oxygenation of FMISO. For the input function the mean value of the VOI data obtained from a large arterial vessel like the descending aorta is used. Besides the VOI based analysis, parametric images are calculated to assess dedicated parameters of the FMISO kinetics.

Besides the compartment analysis a non-compartment model based on the fractal dimension is used. The fractal dimension (FD) is a parameter for the heterogeneity and is calculated for the time activity data of each individual VOI. The values of the fractal dimension vary from 0 to 2 showing the deterministic or chaotic distribution of the tracer activity. We use a subdivision of 7x7 and a maximal SUV of 20 for the calculation of FD.

Functional MRI investigations are performed prior to radiation therapy, at week 5 of radiation therapy and at 6 weeks post treatment. All examinations are performed using a clinical 1.5-T MRI scanner (Magnetom Avanto, Siemens Medical Solutions, Erlangen, Germany).

The standard protocol comprises a coronal and a transversal breath-hold TrueFISP, T2w single-shot half-Fourier TSE (HASTE) and T1w 3D-GRE (VIBE) sequence. Afterwards, a navigator triggered transversal T2w-FatSat sequence (T2-FS BLADE) is performed.

Diffusion weighted imaging is performed using an axial single shot echoplanar (EPI) sequence with and without flow-compensation. A total of ten b-values (0, 10, 25, 50, 100, 200, 300, 400, 500 and 800 s/mm2) is acquired enabling extraction of diffusion and perfusion parameters. DWI parameters are evaluated based on the Intravoxel Incoherent motion (IVIM) model, yielding the parameters perfusion fraction f and diffusion constant D, using in house developed open-source software MITK Diffusion, Version 2011 (downloadable at www.mitk.org). The parameter estimation is based on the assumption that the diffusion measurement is influenced by mainly two effects, a perfusion related effect introduced by the molecules moving in the capillary network (pseudodiffusion coefficient, D*) and extravascular effects of passive diffusion (D). Since a simultaneous nonlinear fit for all parameters D, D*, and the weighting coefficient f can be instable, measurement at b-values greater than 200 s/mm² are used in a first step to estimate f and D as described. D* is then calculated in a second step by using exhaustive search.

Lung cancer perfusion is assessed using a spoiled 3D gradient echo sequence after bolus injection of 0.07 mmol/kg body weight of Gd-DTPA. Ten acquisitions in one expiratory breath hold (10 x 2.25 s = 22 s) are followed by 50 navigator-triggered acquisitions under free breathing. After a co-registration of the 3D data sets, a ROI-based visualization of the signal-time curves is performed.

Furthermore, a time-resolved echoshared gradient echo sequence (TWIST) is performed for assessment of three-dimensional tumor motion (240 x 0.5s = TA 2 min). A dynamic 2D-TrueFISP sequence acquired in coronal orientation crossing the centre of the tumor provides additional information about lung and tumor motion during the breathing cycle.

Contrast-enhanced sequences breath hold 3D-GRE sequence (VIBE) complete this protocol.

The first follow-up is planned 6 weeks post treatment and includes study-related 18F-FMISO dPET-CT and functional MRI examinations. Further regular follow-up visits are scheduled every 3 months for the first 2 years, every 6 months for the following 3 years and thereafter yearly. Individual trial participation is completed three years after patient enrolment or death of the patient.

The therapeutic efficacy will be evaluated through thoracic CT-scan at follow up visits.

The study is a prospective and non-randomized trial with inclusion of 15 patients. Repeated examinations with 18F-FMISO dPET-CT and functional MRI lead to longitudinal data for every patient. The data consists of maps obtained from both measurement devices. Data are quantitative measurements but may be dichotomized or categorized into more than two classes. For all parameters, differences between the site of local relapse and a selected control region are derived and compaired by paired tests at 5% level.

All analyses are exploratory. A sample size calculation cannot be performed because neither standard deviation of the differences has been estimated before, nor the relevant difference is known. Therefore, the study is a pilot study to generate hypotheses for future research.

In the frame of the radiation therapy planning study, virtual radiation therapy strategies are compared to the radiation therapy administered to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Documented inoperable, histologically confirmed NSCLC stage III
* Sufficient remaining lung function (FeV1>1.5 l/s or at least 50 % of the respective individual norm value)
* Karnofsky Performance Score of 70 % or higher.
* Patients > 18 years of age.
* Adequate haematological function (wbc>3000 x 10^3 /ml, thc >100 ×10^6 /ml, Hb>10 g/dl)
* Adequate hepatic and renal function
* Written informed consent

Exclusion Criteria:

* Patient refusal
* Severe concurrent systemic disease
* Claustrophobia
* Cardiac pacemaker
* Other malignancies
* Hypersensitivity to x-ray contrast medium or 18F-FMISO
* Severe renal or hepatic insufficiency
* NSCLC stage I, II or IV
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Standard uptake value (SUV) of 18F-FMISO and k1 and k2 parameters | 3 months
  Primary aim of the study is to assess the correlation between measurements of the standard uptake value (SUV) of 18F-FMISO, as well as measurements of the parameters k1 and k2, which reflect the influx and efflux of FMISO into and out of the cells with functional MRI parameters, such as diffusion coefficients in matched regions of interest in patients with stage III NSCLC treated with intensity modulated radiation therapy (IMRT).

SECONDARY OUTCOMES:
Local recurrence rate | 2 years
  Assessement of the prognostic value of serial 18F-FMISO dPET-CT and functional MRI for 1-year and 2-year local recurrence rate.
Progression free survival | 2 years
  Assessement of the prognostic value of serial 18F-FMISO dPET-CT and functional MRI for 1-year and 2-year progression free survival.
Overall survival | 2 years
  Assessement of the prognostic value of serial 18F-FMISO dPET-CT and functional MRI for overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Debus, Professor, Principal Investigator — University Clinic Heidelberg and German Cancer Research Center
Locations (1):
- German Cancer Research Center, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Askoxylakis V, Dinkel J, Eichinger M, Stieltjes B, Sommer G, Strauss LG, Dimitrakopoulou-Strauss A, Kopp-Schneider A, Haberkorn U, Huber PE, Bischof M, Debus J, Thieke C. Multimodal hypoxia imaging and intensity modulated radiation therapy for unresectable non-small-cell lung cancer: the HIL trial. Radiat Oncol. 2012 Sep 14;7:157. doi: 10.1186/1748-717X-7-157. PMID 22974533